CLINICAL TRIAL: NCT01547754
Title: Inflammation and Function of P-gp in HIV Infection of Brain
Brief Title: Mild Neurocognitive Disorder in HIV Infection of the Brain
Status: Terminated | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 120059; 12-M-0059
Record Dates: First submitted 2012-03-06; First posted 2012-03-08 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2014-08-25

CONDITIONS: HIV-Associated Cognitive Motor Complex
Keywords: Neuroinflammation; HIV; Positron Emission Tomograhy (PET); Mild Neurocognitive Disorder; P-Glycoprotein; Mild Cognitive Disorder; Healthy Volunteer; HV
MeSH Terms: conditions — AIDS Dementia Complex; Neuroinflammatory Diseases; Neurocognitive Disorders

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- Some people with human immunodeficiency virus (HIV) develop problems with thinking and concentration when the virus affects the brain. This is known as mild neurocognitive disorder (MND). Research has shown that some HIV medications do not get through the blood brain barrier very well. P-glycoprotein (P-gp) is a brain protein that is part of the blood brain barrier. Differences in the activity of P-gp may help explain why some people with HIV develop MND. It is also possible that MND is partly due to inflammation in the brain. Researchers want to study P-gp and its effect on MND and HIV infection.

Objectives:

- To study P-gp and brain inflammation related to HIV infection.

Eligibility:

* Individuals between 18 and 60 years of age who have HIV and either do or do not have MND.
* Healthy volunteers between 18 and 60 years of age.

Design:

* Participants will be screened with a medical history and physical exam. Blood and urine samples will be collected.
* Participants will have one outpatient visit and one 3-day inpatient stay.
* At the outpatient visit, participants will provide blood samples and have a lumbar puncture (spinal tap). The spinal tap will collect cerebrospinal fluid for study.
* At the inpatient visit, participants will have two positron emission tomography (PET) scans of the brain. These scans will study brain activity and possible inflammation. One scan will involve a study drug called tariquidar, which blocks the activity of P-gp. A second lumbar puncture will be done before the first PET scan. Blood and urine samples will be collected daily.

DETAILED DESCRIPTION:
Objective:

To determine the relationship among neuroinflammation, Permeability-glycoprotein (P-gp) function and mild neurocognitive disorder (MND), a cognitive disorder associated with HIV infection.

Study Population:

HIV seropositive subjects with MND, HIV seropositive subjects with normal cognitive function, and HIV seronegative control subjects.

Design:

Subjects will undergo history and physical exam, screening laboratory tests, EKG, brain MRI and neuropsychological evaluation. HIV-seropositive subjects will be stratified based on results of neuropsychological evaluation into HIV-seropositive controls (i.e., cognitively normal) and HIV-seropositive with MND. All subjects will receive brain PET imaging with [11C]dLop after P-gp blockade to measure the function of P-gp at the blood-brain barrier. P-gp will be blocked prior to the PET scan with tariquidar. HIV-seropositive subjects will receive one lumbar puncture at baseline and one lumbar puncture after P-gp blockade with tariquidar to measure CSF concentrations of anti-retroviral medications and to measure biomarkers of blood-brain barrier integrity and inflammation in the CSF. HIV-seronegative subjects will receive one lumbar puncture at baseline to measure biomarkers of blood-brain barrier integrity and inflammation in the CSF.

Outcome Measures:

The main outcome measures of the study is brain uptake of [11C]dLop in response to P-gp blockade with tariquidar. We will correct for individual metabolism of tariquidar by measuring the plasma concentration of tariquidar during the P-gp blocked scan.

As a secondary outcome measure, concentrations of anti-retroviral medications in CSF will be measured in HIV seropositive subjects with and without MND. CSF concentrations will be used as a surrogate marker for CNS delivery of anti-retroviral drugs.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Subjects must be between 18 and 60 years of age.
  2. Capable of providing informed consent.
  3. Ambulatory at initial visit.
  4. Speak English fluently
  5. For HIV seropositive subjects:

     1. Confirmation of HIV antibody status by ELISA and Western Blot
     2. Documented HIV-infection for at least one year
     3. On a stable antiretroviral regimen that includes a protease inhibitor for at least 3 months and have a viral load < 400 copies/mL.
     4. Have a primary care physician.

Specific inclusion criteria for mild neurocognitive disorder are as follows:

1. Subject has an acquired mild-to-moderate impairment in cognitive function documented by a score of at least 1 SD below demographically corrected norms on testing of at least two different cognitive domains.
2. The cognitive impairment interferes, at least mildly, with activities of daily living, as determined by neuropsychological interview.
3. The impairment does not meet DSM-IV criteria for delirium or dementia.
4. The impairment is not fully explained by co-morbid conditions.

EXCLUSION CRITERIA:

1. Current Axis I psychiatric illness or severe systemic disease (other than HIV and MND) based on history and physical exam that would make study participation unsafe in the opinion of the investigators.
2. Current alcohol use greater than 14 drinks per week for men and 7 drinks per week for women.
3. Laboratory tests with clinically significant abnormalities. Normal organ and marrow function are defined as: total leukocyte count greater than or equal to 3000 cells/ul, ANC greater than or equal to 1500 cells/ul, platelet count greater than or equal to 100,000 cells/ul, serum creatinine less than or equal to 2.0 times upper limit of normal, hemoglobin greater than or equal to 9.0 g/dL, serum calcium <12.0 mg/dL, AST/ALT less than or equal to 1.5 times the upper limit of normal, PT 1.5 upper limit of normal.
4. EKG finding consistent with ischemic heart disease unless there is documentation of normal cardiac function (e.g., normal stress test or echocardiogram results).
5. Previous research radiation exposure (X-rays, PET scans etc.) that, with the study PET scans, would exceed annual research limits.
6. Pregnancy or breast feeding.
7. Evidence of brain disease such as stroke, tumor, epilepsy, traumatic brain injury, or any neurodegenerative disease on history or on screening MRI.
8. Inability to lay on his/her back for long periods, severe claustrophobia, pacemaker, or other contraindication for MRI.
9. More than moderate hypertension, defined as blood pressure greater than or equal to 160/95 at the time of screening.
10. Current use of illicit drugs based on positive result on urine screen for illicit drugs at the time of screening.
11. Subjects taking medications, other than anti-retroviral drugs, that are known substrates of P-gp that cannot be safely discontinued for this study. Anti-retroviral drugs, particularly protease inhibitors such as ritonavir, that are P-gp substrates are allowed.

Note: The rationale for the exclusion criteria for alcohol use is to avoid alcohol-related cognitive impairment as a confounding factor.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2012-01-09; Study Completion 2014-08-25

PRIMARY OUTCOMES:
Brain uptake of [11C]dLop after pharmacological challenge with the P-gp inhibitor tariquidar.

SECONDARY OUTCOMES:
Cerebrospinal fluid concentrations of antiretroviral drugs and inflammatory markers.

CONTACTS AND LOCATIONS:
Overall Officials: Robert B Innis, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Kaddoumi A, Choi SU, Kinman L, Whittington D, Tsai CC, Ho RJ, Anderson BD, Unadkat JD. Inhibition of P-glycoprotein activity at the primate blood-brain barrier increases the distribution of nelfinavir into the brain but not into the cerebrospinal fluid. Drug Metab Dispos. 2007 Sep;35(9):1459-62. doi: 10.1124/dmd.107.016220. Epub 2007 Jun 25. PMID 17591677
- [Background] Langford D, Grigorian A, Hurford R, Adame A, Ellis RJ, Hansen L, Masliah E. Altered P-glycoprotein expression in AIDS patients with HIV encephalitis. J Neuropathol Exp Neurol. 2004 Oct;63(10):1038-47. doi: 10.1093/jnen/63.10.1038. PMID 15535131
- [Background] Loscher W, Potschka H. Drug resistance in brain diseases and the role of drug efflux transporters. Nat Rev Neurosci. 2005 Aug;6(8):591-602. doi: 10.1038/nrn1728. PMID 16025095